CLINICAL TRIAL: NCT04213859
Title: Emotional Processes During a Randomized Controlled Trial of Virtual Reality Exposure Treatment for Flight Phobia
Brief Title: Emotional Processes in VR Exposure Treatment for Flight Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idan Moshe Aderka (Other)
Responsible Party: Sponsor-Investigator, Idan Moshe Aderka, Ph.D. Senior Lecturer, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6557-19-SMC
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Fear of Flying
MeSH Terms: conditions — Aerophobia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exposure Therapy (VRET) (Experimental): 1. st stage: Participants will receive information about the study, complete measures of fear of flying and emotional variables, and undergo a diagnostic interview for flight phobia and additional disorders.
  2. nd stage: During the week prior to treatment, participants will complete a brief measure of emotion-related variables every evening at a fixed time (08:00 pm).
  3. rd stage: Participants will receive therapy for fear of flying using a Virtual Reality (VR) simulator. Therapy sessions will be held once a week during 4 weeks. Participants will complete a brief measure of emotion-related variables at a random time during the 12 hours before the therapy session at a random time during the 12 hours after the therapy session. This will occur for every therapy session.
  4. th stage: After treatment, participants will complete measures of fear of flying and emotional variables.
  Interventions: Behavioral: VRET - Virtual Reality Exposure Therapy
- control (No Intervention): 1. st stage: Participants will receive information about the study, complete measures of fear of flying and emotional variables, and undergo a diagnostic interview for flight phobia and additional disorders.
  2. nd stage: During five weeks no therapy will be administered. Participants will fill questionnaires as follows: During the first week, participants will complete emotional measures every evening at a fixed time (08:00 pm)
  3. rd stage: During each of the following 4 weeks, participants will complete two emotional measures during a 24 hour period.
  4. th stage: Participants will complete measures of fear of flying and emotional variables.

INTERVENTIONS:
Behavioral: VRET - Virtual Reality Exposure Therapy — VRET will include 4 weekly 1-hour sessions over the course of 4 weeks. The treatment protocol is based on the Virtual Reality (VR) treatment manual guidelines (Rothbaum & Hodges, 1997,1999) and includes psychoeducation, anxiety management training, cognitive restructuring and exposure. The first therapy session focuses on creating an individually-tailored conceptualization and treatment plan. Following this process, participant and therapist conduct a short introductory VR flight exposure simulation to familiarize the participant with the VRET apparatus. The VRET apparatus is an advanced, large-scale VR system that allows maximal immersion within the virtual environment. The second, third and fourth sessions include psychoeducation, relaxation training, cognitive restructuring and individually-tailored VR exposures (the therapist can manipulate the turbulence level and other flight-related variables to fit participants' fears and current progress).
  Arms: Virtual Reality Exposure Therapy (VRET)

SUMMARY:
This study will assess emotional processes and their relation to treatment outcomes during Virtual reality exposure therapy for Flight Phobia. The researchers hypothesize treatment outcomes will be associated with positive changes in emotional constructs

DETAILED DESCRIPTION:
Emotional constructs and emotion regulation capacities play a central role in the severity of anxiety disorders and are directly related to treatment outcomes in different anxiety disorders. In this study we will examine the relation between positive and negative affect, emotion regulation, emotional instability, emotional differentiation, experiential avoidance and therapy outcomes in participants undergoing Virtual Reality Exposure Therapy for Flight Phobia. We assume that treatment outcomes will be positively related to changes in the regulation, management and experience of emotions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Flight phobia based on a structured interview
* possession of a smartphone with an active data plan

Exclusion Criteria:

* cardiovascular disease
* neurological disorders and history of epilepsy
* psychosis
* major depression
* suicidal behavior
* substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in FAS (Flight Anxiety Situations Questionnaire) scores | Two weeks prior to therapy and one week after last therapy session (therapy includes 4 weekly 1-hour sessions over the course of 4 weeks)
  The Flight Anxiety Situations Questionnaire (Van Grewen, Spinhoven, Van-Dyck, & Dikstra, 1999) is a 32-item, 5-point Likert-scale (1= no anxiety to 5=overwhelming anxiety). The FAS evaluates flight-related anxiety in various situations and includes 3 factors: generalized, anticipatory and in-flight anxiety.
Changes in FAM (Flight Anxiety Modality questionnaire) scores | Two weeks prior to therapy and one week after last therapy session (therapy includes 4 weekly 1-hour sessions over the course of 4 weeks).
  The Flight Anxiety Modality (FAM) questionnaire (Van Grewen et al. 1999) assesses somatic and cognitive aspects of Flight Phobia. It includes 18 items that are rated using a 5-point scale (1=not at all, 5=very intensely). The somatic factor assesses physiological symptoms and the cognitive factor assesses anxiety-provoking cognitions

CONTACTS AND LOCATIONS:
Overall Officials: Asaf Caspi, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No